CLINICAL TRIAL: NCT03213262
Title: Is Anxiety Affect the Anesthesia Type Performed In Patients During Caeserean Section ?
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assist.Prof., Tokat Gaziosmanpasa University
Other Study IDs: 17-KAEK-076
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anesthesia: The effect of anxiety on the choice of anesthesia will be evaluated.
- spinal anesthesia: Cesarean patients with spinal anesthesia

SUMMARY:
In this study, investigators wanted to investigate the effect of preoperative anxiety level on anesthesia preference of patient. Before surgery, patients will fill the forms of Pain catastrophising scale (PCS), Beck depression and Beck anxiety scale. After surgery, these forms will be evaluated according to the choice of anesthesia.

DETAILED DESCRIPTION:
Anxiety is present due to many gait in the preoperative period. In studies that investigated anxiety levels in the preoperative period was found that 60-80% of the patients had significant anxiety. The present study is aimed to investigate the effect of preoperative anxiety level on anesthesia preference of cesarean patients. After approval, patients enrolled in the study is invited to complete the Pain Catastrophizing Scale questionnaire, Beck depression and Beck anxiety scale. After surgery, The effect of anxiety on the choice of anesthesia will be evaluated (general or spinal anesthesia).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years
* Planned to undergo ceserean
* An American Society of Anesthesiologists score of 1 or 2

Exclusion Criteria:

* Psychiatric diseases
* Rejected to participation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ceserean patients
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-24 (Actual)

PRIMARY OUTCOMES:
Anesthesia preference and anxiety | one time in three months
  The spinal and general anesthesia preference according to the anxiety level of cesarean patients

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Principal Investigator — Gaziosmanpasa university
Locations (1):
- Gaziosmanpasa university, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No